CLINICAL TRIAL: NCT01454570
Title: The ReWalk Exoskeletal Walking System for Persons With Paraplegia
Acronym: VA_ReWalk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ann M. Spungen, EdD, Associate Director of CoE / Health Science Specialist, James J. Peters Veterans Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: JJPVAMC: SPU-09-11; Protocol#: SPU-09-11 (Other: JamesJPetersVAMC)
Record Dates: First submitted 2011-09-14; First posted 2011-10-19 (Estimated); Results first posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Paraplegia
Keywords: exoskeleton walking system; paraplegia; paralysis
MeSH Terms: conditions — Paraplegia; Paralysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Powered Exoskeleton (Experimental): persons with SCI trained to use a powered exoskeleton to ambulate overground
  Interventions: Device: powered exoskeleton

INTERVENTIONS:
Device: powered exoskeleton

SUMMARY:
It is well appreciated that an extreme sedentary lifestyle from paralysis, contributes to many secondary medical problems such as diabetes and insulin resistance, obesity, constipation, poor blood pressure regulation, cardiovascular disease, reduced quality of life, and more. The ReWalk-I exoskeleton walking device permits investigation of the potential benefits of frequent upright posture and walking on many of the secondary consequences of spinal cord injury. The researchers are investigating the ability of persons with paraplegia to learn to stand and walk with the ReWalk-I and the effects of being upright and walking on several of these secondary medical consequences of spinal cord injury.

DETAILED DESCRIPTION:
Potential participants will be pre-screened with the inclusion criteria for eligibility. The informed consent process will begin for those participants who have been determined to meet the inclusion criteria. After the potential participant's signed consent has been provided, further evaluations for eligibility will be performed (e.g., there are several medical and physical exclusion criteria). Those potential participants who meet both the inclusion and exclusion criteria will be eligible to enroll into the ReWalk-I study. Baseline evaluations and personalized measurements for fitting to the ReWalk-I will be performed over one week, before the training sessions begin. The ReWalk sessions will consist of a Learning Phase (12 sessions in 4 weeks) and a Training Phase (18 sessions in 6 weeks). These times may vary by each participant's ReWalk learning curve. Training will begin with sit-to-stand, stand-to-sit, and standing balance activities. Progression to walking will occur as skills advance. Each session will be an average 50 minutes, with 3 sessions per week. The skills to be learned include 1) sit-to-stand, 2) stand-to-sit, 3) 2-arm standing balance, 4) 1-arm standing balance, 5) walking, and 6) stair climbing. The study evaluations will be repeated after the Learning Phase, after the Training Phase and 1-month post training follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females with paraplegia
2. Duration of SCI >6 months
3. Ages 18 to 65 y
4. Height 160 to 190cm (63-75in or 5'3" to 6'3")
5. Weight <100kg (<220 lb)
6. Ability to give informed consent

Exclusion Criteria:

1. Diagnosis of neurological injury other than SCI including:

   * Multiple sclerosis (MS)
   * Stroke
   * Cerebral Palsy (CP)
   * Amyotrophic lateral sclerosis (ALS)
   * Traumatic Brain injury (TBI)
   * Spina bifida
   * Parkinson's disease (PD)
   * Other neurological condition that the study physician considers in his/her clinical judgment to be exclusionary
2. Severe concurrent medical disease, illness or condition
3. Recent lower extremity fracture within the past 2 years;
4. DXA results indicating a t-score below -3.0 and knee BMD <0.70 gm/cm2
5. Systemic or peripheral infection
6. Atherosclerosis, congestive heart failure, or history of myocardial infarction
7. Trunk and/or lower extremity pressure ulcers;
8. Other illness, that the study physician considers in his/her clinical judgment to be exclusionary
9. Severe spasticity (defined by an Ashworth score of >4.0 or clinical impression of the study physician or physical therapist)
10. Significant contractures defined as flexion contracture limited to 35º at the hip and 20º at the knee;
11. Diagnosis of heterotrophic ossification of the lower extremities;
12. Femoral neck or the total proximal femur bone mineral density T-scores < -3.0
13. Psychopathology documentation in the medical record or history of that may conflict with study objectives
14. Hypertension (SBP>140, DBP>90)
15. Pregnancy and/or lactating females

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-02; Primary Completion 2015-08-08 (Actual); Study Completion 2015-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann M Spungen, EdD, Principal Investigator — Bronx JJPVAMC CoE 7A-13
Locations (1):
- James J. Peters Veterans Affairs Medical Center; Center of Excellence for the Major Consequences of SCI., The Bronx, New York, United States

REFERENCES:
- [Derived] Tsai CY, Asselin PK, Hong E, Knezevic S, Kornfeld SD, Harel NY, Spungen AM. Exoskeletal-assisted walking may improve seated balance in persons with chronic spinal cord injury: a pilot study. Spinal Cord Ser Cases. 2021 Mar 12;7(1):20. doi: 10.1038/s41394-021-00384-8. PMID 33712561
- [Derived] Asselin P, Cirnigliaro CM, Kornfeld S, Knezevic S, Lackow R, Elliott M, Bauman WA, Spungen AM. Effect of Exoskeletal-Assisted Walking on Soft Tissue Body Composition in Persons With Spinal Cord Injury. Arch Phys Med Rehabil. 2021 Feb;102(2):196-202. doi: 10.1016/j.apmr.2020.07.018. Epub 2020 Nov 7. PMID 33171129
- [Derived] Asselin P, Knezevic S, Kornfeld S, Cirnigliaro C, Agranova-Breyter I, Bauman WA, Spungen AM. Heart rate and oxygen demand of powered exoskeleton-assisted walking in persons with paraplegia. J Rehabil Res Dev. 2015;52(2):147-58. doi: 10.1682/JRRD.2014.02.0060. PMID 26230182
- See also: A Study Testing Safety and Tolerance of the ReWalk Exoskeleton Suit (RW) — http://clinicaltrials.gov/ct2/show/NCT00627107

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited, consented, screened and eligible subjects were enrolled at the James J Peters VAMC
Groups:
- Exoskeleton: Participants trained to use powered exoskeleton for overground ambulation.
Period: Overall Study
Arm/Group | Exoskeleton
Started | 19
Completed | 10
Not Completed | 9
Not completed — Withdrawal by Subject | 2
Not completed — Screen Failure | 7

BASELINE CHARACTERISTICS:
Groups:
- Exoskeleton: Trained to use powered exoskeleton for overground ambulation
Arm/Group | Exoskeleton
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Count to Achieve Mobility Skills
Description: 1. To determine efficacy for mobility defined as the ability to perform the following with the ReWalk-I exoskeletal system, without staff assistance:
  1. Sit-to-stand,
  2. Stand-to-sit,
  3. Standing balance for 1 minutes with both crutches,
  4. Standing balance for 30 seconds with one crutch,
  5. Ten meter walk in ≤2 minutes,
  6. Walk ≥30 meters in 6-minutes, and
  7. Ascend, turn around and descend 4 stairs in 5 minutes.
Time Frame: ReWalk training at 4 and 12 weeks, and 1-month follow-up
Population: number of participants that were able to achieve the mile stone described in outcome measure description
Measure: Count of Participants; unit: Participants
Arm/Group | Exoskeleton
Number analyzed (Participants) | 12
Participants
  No assistance sit-to-stand (4 weeks): Passed | 9
  No assistance sit-to-stand (4 weeks): Not Passed | 3
  No assistance sit-to-stand (4 weeks): Not Tested | 0
  No assistance sit-to-stand (12 weeks): Passed | 10
  No assistance sit-to-stand (12 weeks): Not Passed | 1
  No assistance sit-to-stand (12 weeks): Not Tested | 1
  No assistance sit-to-stand (1 month follow-up): Passed | 9
  No assistance sit-to-stand (1 month follow-up): Not Passed | 1
  No assistance sit-to-stand (1 month follow-up): Not Tested | 2
  No assistance stand-to-sit (4 week): Passed | 9
  No assistance stand-to-sit (4 week): Not Passed | 3
  No assistance stand-to-sit (4 week): Not Tested | 0
  No assistance stand-to-sit (12 week): Passed | 10
  No assistance stand-to-sit (12 week): Not Passed | 1
  No assistance stand-to-sit (12 week): Not Tested | 1
  No assistance stand-to-sit (1 month follow-up): Passed | 9
  No assistance stand-to-sit (1 month follow-up): Not Passed | 1
  No assistance stand-to-sit (1 month follow-up): Not Tested | 2
  No assist standing 2 crutches 1 min (4 weeks): Passed | 11
  No assist standing 2 crutches 1 min (4 weeks): Not Passed | 1
  No assist standing 2 crutches 1 min (4 weeks): Not Tested | 0
  No assist standing 2 crutches 1 min (12 weeks): Passed | 11
  No assist standing 2 crutches 1 min (12 weeks): Not Passed | 1
  No assist standing 2 crutches 1 min (12 weeks): Not Tested | 0
  No assist standing 2 crutches 1 min (1 mo FU): Passed | 11
  No assist standing 2 crutches 1 min (1 mo FU): Not Passed | 0
  No assist standing 2 crutches 1 min (1 mo FU): Not Tested | 1
  No assist standing 1 crutch 30 sec (4 weeks): Passed | 10
  No assist standing 1 crutch 30 sec (4 weeks): Not Passed | 2
  No assist standing 1 crutch 30 sec (4 weeks): Not Tested | 0
  No assist standing 1 crutch 30 sec (12 weeks): Passed | 11
  No assist standing 1 crutch 30 sec (12 weeks): Not Passed | 0
  No assist standing 1 crutch 30 sec (12 weeks): Not Tested | 1
  No assist standing 1 crutch 30 sec (1 mo FU): Passed | 10
  No assist standing 1 crutch 30 sec (1 mo FU): Not Passed | 0
  No assist standing 1 crutch 30 sec (1 mo FU): Not Tested | 2
  No assistance 10 walk in ≤2 min (4 weeks): Passed | 4
  No assistance 10 walk in ≤2 min (4 weeks): Not Passed | 8
  No assistance 10 walk in ≤2 min (4 weeks): Not Tested | 0
  No assistance 10 walk in ≤2 min (12 weeks): Passed | 7
  No assistance 10 walk in ≤2 min (12 weeks): Not Passed | 4
  No assistance 10 walk in ≤2 min (12 weeks): Not Tested | 1
  No assistance 10 walk in ≤2 min (1 mo FU): Passed | 6
  No assistance 10 walk in ≤2 min (1 mo FU): Not Passed | 4
  No assistance 10 walk in ≤2 min (1 mo FU): Not Tested | 2
  No assistance walk ≥30 meters in 6-min (4 weeks): Passed | 4
  No assistance walk ≥30 meters in 6-min (4 weeks): Not Passed | 8
  No assistance walk ≥30 meters in 6-min (4 weeks): Not Tested | 0
  No assistance walk ≥30 meters in 6-min (12 weeks): Passed | 7
  No assistance walk ≥30 meters in 6-min (12 weeks): Not Passed | 4
  No assistance walk ≥30 meters in 6-min (12 weeks): Not Tested | 1
  No assistance walk ≥30 meters in 6-min (1 mo FU): Passed | 6
  No assistance walk ≥30 meters in 6-min (1 mo FU): Not Passed | 4
  No assistance walk ≥30 meters in 6-min (1 mo FU): Not Tested | 2
  No assistance ascend and descend stairs (4 weeks): Passed | 1
  No assistance ascend and descend stairs (4 weeks): Not Passed | 3
  No assistance ascend and descend stairs (4 weeks): Not Tested | 8
  No assistance ascend and descend stairs (12 weeks): Passed | 4
  No assistance ascend and descend stairs (12 weeks): Not Passed | 0
  No assistance ascend and descend stairs (12 weeks): Not Tested | 8
  No assistance ascend and descend stairs (1 mo FU): Passed | 4
  No assistance ascend and descend stairs (1 mo FU): Not Passed | 0
  No assistance ascend and descend stairs (1 mo FU): Not Tested | 8

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Exoskeleton
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 7/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exoskeleton (N=12)
Skin Abrasion / bruising /redness (Skin and subcutaneous tissue disorders) | 1 (1)
Skin abrasion (Skin and subcutaneous tissue disorders) | 1 (1) — Lower Back Abraision
R Medial Malleolus Redness (Skin and subcutaneous tissue disorders) | 1 (1) — Skin Abraision / bruising /redness
L Lateral Malleolus Skin Abraision (Skin and subcutaneous tissue disorders) | 1 (1) — Skin Abrasion / bruising /redness
Tailbone Skin Breakdown (Skin and subcutaneous tissue disorders) | 1 (1) — Skin Abrasion/ bruising /redness
R Ischial Area Abasion (Skin and subcutaneous tissue disorders) | 1 (1) — Skin Abrasion / bruising /redness
L Medial Malleolus Abrasion (Skin and subcutaneous tissue disorders) | 1 (1) — Skin Abrasion / bruising /redness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes